CLINICAL TRIAL: NCT00466466
Title: A Phase Ib Study Investigating the Combination of RAD001 With Cisplatin and Etoposide in Patients With Extensive-stage Small-cell Lung Cancer Not Previously Treated With Chemotherapy
Brief Title: Safety of RAD001 in Combination With Cisplatin and Etoposide in Lung Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2116
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2011-11

CONDITIONS: Small-Cell Lung Cancer
Keywords: Small-Cell Lung Cancer; SCLC; Advanced Lung Cancer; RAD; RAD001; Chemotherapy; Cisplatin; Etoposide
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Everolimus

ARMS (2):
- Daily dosing RAD001 (Experimental)
  Interventions: Drug: Everolimus
- Weekly dosing RAD001 (Experimental)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — RAD001 will be supplied by Novartis as tablets in 3 different dosage strengths, 2.5, 5 and 10 mg. The drug will be packaged in blisters containing 10 tablets per blister. Blisters and packaging will be compliant with local regulations and be printed in local language.
  Other Names: RAD001

SUMMARY:
This study aims to establish a tolerable dose level and regimen of RAD001 in combination with cisplatin and etoposide (standard-of-care chemotherapy) in patients with extensive stage small-cell lung cancer (SCLC) who have not previously been treated with systemic chemotherapy.

ELIGIBILITY:
Inclusion criteria:

* Patients with histologically or cytologically confirmed diagnosis of extensive disease small-cell lung cancer (ED SCLC)
* Age ≥ 18 years
* WHO Performance Status Grade ≤ 1 (ie. ability to perform normal daily functions)
* Adequate bone marrow, liver and renal function

Exclusion criteria:

* Chronic steroid treatment
* Prior treatment with chemotherapy for advanced lung cancer
* Prior treatment with mTOR inhibitors
* Active bleeding conditions, skin conditions, gastrointestinal disorders, mouth ulcers, eye conditions, chronic liver or kidney disorders, uncontrolled diabetes, infections or other severe medical conditions
* Symptomatic or uncontrolled brain metastases
* Other cancers within the past 5 years
* Pregnant or breastfeeding women

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-04; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) rate will be measured at End-of-Cycle 1 | Day 21

SECONDARY OUTCOMES:
Relative dose intensity (RDI) of carboplatin and paclitaxel will be evaluated upon completion of the dose escalation within each regimen | within 6 cycles (Day 126)
PK parameters derived from the PK profile of treatment drugs when administered alone or in combination will be evaluated during the first 6 cycles | During the first 6 cycles
Overall tumor response | Every 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (5):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas
  - Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas
- Novartis Investigative Site, Paris, France

REFERENCES:
- See also: Results for CRAD001C2116 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4726